CLINICAL TRIAL: NCT00043147
Title: A Phase III, Randomized, Placebo-Controlled, Multicenter Study of the Safety, Efficacy, and Pharmacokinetics of Oral Beclomethasone 17, 21-Dipropionate (BDP) in Conjunction With Ten Days of High-Dose Prednisone Therapy in the Treatment of Patients With Grade II Graft vs. Host Disease With Gastrointestinal Symptoms
Brief Title: Beclomethasone Plus Prednisone in Treating Patients With Graft-Versus-Host Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: ENTERON-00-02; MSKCC-01149; CDR0000256305 (Registry Identifier: PDQ (Physician Data Query)); NCI-G02-2098; RPCI-DS-01-09
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2004-12

CONDITIONS: Graft Versus Host Disease
Keywords: graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Beclomethasone; Methylprednisolone; Prednisone

INTERVENTIONS:
Drug: beclomethasone dipropionate
Drug: methylprednisolone
Drug: prednisone

SUMMARY:
RATIONALE: Beclomethasone combined with prednisone may be an effective treatment for graft-versus-host disease caused by stem cell transplantation. It is not yet known if prednisone is more effective with or without beclomethasone in treating gastrointestinal graft-versus-host disease.

PURPOSE: Randomized phase III trial to determine the effectiveness of prednisone with or without beclomethasone in treating patients who have graft-versus-host disease afftecting the gastrointestinal system.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of beclomethasone dipropionate and prednisone vs placebo and prednisone, in terms of time to treatment failure, in patients with grade II graft-vs-host disease with gastrointestinal symptoms.
* Compare the proportion of treatment failures on study days 10, 30, 50, 60, and 80 in patients treated with these regimens.
* Compare the cumulative systemic corticosteroid exposure in patients treated with these regimens.
* Compare the incidence and degree of hypothalamic-pituitary-adrenal axis suppression in patients treated with these regimens who have not experienced treatment failure by study day 50.
* Compare the safety of these regimens in these patients.
* Compare the total deaths and causes of death through 200 days post-transplantation of patients treated with these regimens.
* Assess the pharmacokinetic profile of beclomethasone dipropionate in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, parallel, multicenter study. Patients are stratified according to graft tissue source (2 HLA haplotype-identical sibling vs all others) and topical steroid use at baseline (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral beclomethasone dipropionate 4 times daily on days 1-50. Patients also receive oral prednisone (or methylprednisolone IV) twice daily on days 1-10 with a rapid taper on days 11-17 followed by low-dose prednisone on days 18-80.
* Arm II: Patients receive oral placebo 4 times daily on days 1-50. Patients also receive prednisone (or methylprednisolone) as in arm I.

In both arms, treatment continues in the absence of poorly controlled GVHD at day 10 or unacceptable toxicity.

Patients are followed at days 51, 60, and 80 and then at 200 days post-transplantation.

PROJECTED ACCRUAL: A total of 130 patients (65 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed graft-vs-host disease (GVHD) with gastrointestinal symptoms

  * Endoscopic evidence of grade II intestinal GVHD without another plausible etiology
  * Confirmed by biopsy of colon, stomach, small intestine, esophagus, or skin within 72 hours prior to study entry
* At least 10 days post allogeneic hematopoietic stem cell transplantation
* Received prior anti-candidal prophylaxis of the oropharynx with an effective drug
* Confirmed absence of intestinal infection within the past 7 days
* No liver GVHD with bilirubin greater than 3 mg/dL
* No skin GVHD other than a slowly evolving rash that involves no more than 50% of the body surface
* No more than 1,000 mL/day of diarrhea on any 1 day within the past 3 days

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Not specified

Life expectancy

* At least 3 months

Hematopoietic

* Not specified

Hepatic

* See Disease Characteristics

Renal

* Not specified

Other

* HIV negative
* Able to swallow tablets
* No multi-organ failure
* No sepsis syndrome
* No other condition with high mortality
* No infection of the mouth or esophagus with a fungal organism
* No persistent vomiting of oral intake
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 30 days since prior biologic agents

Chemotherapy

* Not specified

Endocrine therapy

* At least 30 days since prior systemic (oral or parenteral) prescription corticosteroids administered for prophylaxis or treatment of GVHD or another inflammatory disease process
* Concurrent dexamethasone as an antiemetic or to lessen side effects during medication or blood product administration allowed

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Other

* No prior beclomethasone dipropionate
* At least 30 days since prior investigational drugs or devices
* Concurrent immunosuppressants (e.g., cyclosporine, tacrolimus, sirolimus, methotrexate, or mycophenolate mofetil) allowed for GVHD prophylaxis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-04; Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel-Angel Perales, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York